CLINICAL TRIAL: NCT02594163
Title: A Randomized, Open Label, Phase 2 Study of Rituximab and Bendamustine With or Without Brentuximab Vedotin for Relapsed or Refractory CD30-Positive Diffuse Large B-Cell Lymphoma
Brief Title: Study of Rituximab and Bendamustine With or Without Brentuximab Vedotin for CD30 Positive Diffuse Large B-cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision based on portfolio prioritization
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGN35-023
Record Dates: First submitted 2015-10-30; First posted 2015-11-02 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Diffuse Large B-cell Lymphoma Refractory; Follicular B-cell Non-Hodgkin's Lymphoma
MeSH Terms: interventions — Brentuximab Vedotin; Rituximab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brentuximab Vedotin (Experimental): Subjects randomized to the brentuximab vedotin arm will receive IV infusions of brentuximab vedotin followed by bendamustine on day 1, and rituximab followed by bendamustine on day 2 of each 21 day cycle.
  Interventions: Drug: Brentuximab Vedotin; Drug: Rituximab; Drug: Bendamustine
- Rituximab,Bendamustine control (Active Comparator): Subjects randomized to the control arm will receive IV infusions of rituximab on day 1 or day 2 and bendamustine on both days 1 and 2 of each 21 day cycle.
  Interventions: Drug: Rituximab; Drug: Bendamustine

INTERVENTIONS:
Drug: Brentuximab Vedotin
  Other Names: Adcetris
  Arms: Brentuximab Vedotin
Drug: Rituximab
  Other Names: Rituxan
Drug: Bendamustine
  Other Names: Treanda

SUMMARY:
This is a randomized, open-label, multicenter, Phase 2 clinical trial designed to evaluate the efficacy and safety of brentuximab vedotin in combination with rituximab and bendamustine for the treatment of patients with relapsed or refractory CD30-positive diffuse large B-cell lymphoma (DLBCL) after failure of second-line salvage therapy or as second-line treatment in patients ineligible for autologous stem cell transplant (ASCT).

DETAILED DESCRIPTION:
Patients will be randomized in a 1:1 manner to receive rituximab plus bendamustine with or without brentuximab vedotin. Patients who respond to combination treatment containing brentuximab vedotin and do not experience excessive toxicity may receive additional single-agent brentuximab vedotin following combination treatment, for up to an additional 10 cycles (up to 16 total cycles of treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed CD30-positive DLBCL or grade 3b follicular non-Hodgkin lymphoma (NHL).
2. Patients must have relapsed or refractory disease following:

   1. second-line or greater salvage systemic therapy, or
   2. frontline cytotoxic systemic therapy, for patients who are ineligible for stem cell transplant (SCT).
3. Age 18 years and older.
4. Fluorodeoxyglucose (FDG)-avid disease by positron emission tomography (PET).
5. An Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.
6. Acceptable blood test results.
7. Females of childbearing potential must have a negative pregnancy test result within 7 days prior to the first dose of study drug.
8. Females of childbearing potential and males who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 6 months following the last dose of brentuximab vedotin or 12 months following the last dose of rituximab, whichever is later.
9. Patients must provide written informed consent.

Exclusion Criteria:

1. History of another invasive malignancy that has not been in remission for at least 1 year. (Exceptions are nonmelanoma skin cancer, curatively treated localized prostate cancer, ductal carcinoma, and cervical carcinoma or a squamous intraepithelial lesion on PAP smear).
2. History of progressive multifocal leukoencephalopathy (PML).
3. Cerebral/meningeal disease related to the underlying malignancy, unless definitively treated.
4. Viral, bacterial, or fungal infection within 2 weeks prior to the first dose of treatment.
5. Chemotherapy, radiotherapy, biologics, and/or other antitumor treatment with immunotherapy that is not completed 4 weeks prior to first dose of study drug.
6. Females who are pregnant or breastfeeding.
7. Known allergy to any study drug or ingredient contained in the drug formulation of any of the study drugs.
8. Known to be positive for hepatitis B. Known to have active hepatitis C infection or on antiviral therapy for hepatitis C within the last 6 months.
9. Known to be positive for human immunodeficiency virus (HIV).
10. Patients with previous allogeneic stem cell transplant.
11. Previous treatment with brentuximab vedotin or bendamustine.
12. Intolerable toxicity to prior rituximab therapy.
13. Current therapy with other investigational agents.
14. Lung disease unrelated to underlying malignancy.
15. History of a stroke or transient ischemic attack, unstable angina, myocardial infarction, or cardiac symptoms within 6 months prior to the first dose of treatment.
16. Congestive heart failure.
17. Significant peripheral sensory or motor neuropathy at the start of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-10; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Manley, MD, Study Director — Seagen Inc.
Locations (50):
- United States (22):
  - City of Hope, Duarte, California
  - Sansum Clinic - West Pueblo, Santa Barbara, California
  - Good Samaritan Hospital, Torrance, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - Rocky Mountain Cancer Center, Aurora, Colorado
  - Kaiser Permanente Oncology, Lonetree, Colorado
  - Illinois Cancer Specialists, Niles, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Saint Francis Cancer Treatment Center, Grand Island, Nebraska
  - Hematology and Oncology Associates of Northern New Jersey, P.A., Morristown, New Jersey
  - Willamette Valley Cancer Institute and Research Center, Springfield, Oregon
  - Bon Secours Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Institutional Review Board, Greenville, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Oncology - Flower Mound, Denton, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - Virginia Mason Clinical Research, Seattle, Washington
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
- Czechia (3):
  - FN Brno, Brno
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Fakultní nemocnice Královské Vinohrady, Prague
- France (9):
  - Centre Hospitalier Regional Universitaire (CHRU) Brest - Hopital Morvan, Brest
  - CHU Côte de Nacre - Caen, Caen
  - Centre Hospitalier des Oudairies, La Roche-sur-Yon
  - Centre Hospitalier du Mans, Le Rocher
  - CHR Metz, Metz
  - Centre Hospitalier Universitaire de Nantes (CHU Nantes) - Hotel Dieu, Nantes
  - Centre Hospitalier de Perpignan, Perpignan
  - Centre Hospitalier Universitaire (CHU) de Poitier- Hopital de la Miletrie - Hopital Jean Bernard, Poitiers
  - Centre Hospitalier Universitaire de Rennes, Hôpital Pontchaillou, Rennes
- Italy (6):
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico S.Orsola-Malpighi, Bologna
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - IRCSS Policlinico San Matteo, Pavia
  - Azienda Policlinico Umberto I di Roma, Roma
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - A.O Ospadale Di Circolo E Fondazione Macchi, Varese
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Wojewódzki Szpital Specjalistyczny, Lodz
- Spain (4):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Hospital Universitario La Fe, Valencia
  - Hospital Clinico Universitario Lozano Blesa de Zaragoza, Zaragoza
- United Kingdom (4):
  - University Hospital's Birmingham NHS Foundation trust-Queen Elizabeth Hospital, Birmingham
  - Liverpool and Broadgreen Hospital, Liverpool
  - Maidstone and Tunbridge Wells NHS Trust, Maidstone
  - Christie Hospital NHS Foundation Trust, Manchester

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab, Bendamustine Control: Subjects randomized to the control arm will receive IV infusions of rituximab on day 1 or day 2 and bendamustine on both days 1 and 2 of each 21 day cycle.
  Rituximab
  Bendamustine
- Brentuximab Vedotin Plus Rituximab Plus Bendamustine: Subjects randomized to the brentuximab vedotin arm will receive IV infusions of brentuximab vedotin followed by bendamustine on day 1, and rituximab followed by bendamustine on day 2 of each 21 day cycle.
  Brentuximab Vedotin
  Rituximab
  Bendamustine
Period: Treatment Period
Arm/Group | Rituximab, Bendamustine Control | Brentuximab Vedotin Plus Rituximab Plus Bendamustine
Started | 12 | 13
Completed | 5 | 1
Not Completed | 7 | 12
Not completed — Progressive disease | 2 | 3
Not completed — Adverse Event | 1 | 5
Not completed — Physician Decision | 1 | 3
Not completed — Study termination by sponsor | 2 | 1
Not completed — Other, Non-AE | 1 | 0
Period: Follow-up Period
Arm/Group | Rituximab, Bendamustine Control | Brentuximab Vedotin Plus Rituximab Plus Bendamustine
Started | 12 (All participants were to be followed after treatment) | 13 (All participants were to be followed after treatment)
Completed | 1 | 1
Not Completed | 11 | 12
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Study Termination by Sponsor | 6 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 2 | 5
Not completed — Adverse Event | 0 | 1
Not completed — Progressive Disease | 2 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab, Bendamustine Control | Brentuximab Vedotin Plus Rituximab Plus Bendamustine | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 10
  >=65 years | 6 | 9 | 15
Age, Continuous [Median (Full Range); unit: years] | 64.5 [47 to 85] | 68.0 [40 to 79] | 68.0 [40 to 85]
Sex: Female, Male [Count of Participants; unit: Participants] — According to programmed outputs, 7 patients in the R+B comparator arm were female (sex data were missing for 1 patient). Upon review of available data in a case report form, it was discovered the patient's sex was reported to be female. Therefore 8 patients in the R+B arm are female, a noted discrepancy between the CSR.
  Participants
    Female | 8 | 6 | 14
    Male | 4 | 7 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 7 | 10 | 17
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 11 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5
  Czechia | 1 | 0 | 1
  Poland | 1 | 0 | 1
  Italy | 3 | 4 | 7
  United Kingdom | 1 | 4 | 5
  France | 4 | 2 | 6
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Measure Description: 0=Normal activity; 1=Symptoms but ambulatory; 2=In bed <50% of the time; 3= In bed >50% of the time; 4=100% bedridden; 5=Dead
  Participants
    0: Normal Activity | 7 | 6 | 13
    1: Symptoms but ambulatory | 5 | 4 | 9
    2: In bed less than 50% of the time | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of patients who achieve a Complete Response (CR) (including Complete Metabolic Response (CMR)) or Partial Response (PR) (including Partial Metabolic Response (PMR)) as best response to combination therapy on study
Time Frame: Approximately 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab, Bendamustine Control | Brentuximab Vedotin Plus Rituximab Plus Bendamustine
Number analyzed (Participants) | 12 | 13
percentage of participants | 91.7 [61.5 to 99.8] | 61.5 [31.6 to 86.1]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from randomization to disease progression/relapse, receipt of subsequent lymphoma chemotherapy other than the components of the study treatment regimen, or death from any cause, whichever occurs first.
Time Frame: Up to 11.8 months
Measure: Median (Full Range); unit: months
Arm/Group | Rituximab, Bendamustine Control | Brentuximab Vedotin Plus Rituximab Plus Bendamustine
Number analyzed (Participants) | 12 | 13
months | 4.9 [1.6 to 11.8] | 3.7 [0.8 to 11.5]

3. Secondary Outcome: Complete Remission (CR) Rate
Description: CRR is the proportion of patients who achieve CR (including Complete Metabolic Response (CMR)) as best response to combination therapy on study.
Time Frame: Approximately 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab, Bendamustine Control | Brentuximab Vedotin Plus Rituximab Plus Bendamustine
Number analyzed (Participants) | 12 | 13
Participants | 8 | 7

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from first observation of response to disease progression/relapse, receipt of subsequent lymphoma chemotherapy other than the components of the study treatment regimen, or death from any cause, whichever occurs first.
Time Frame: Up to 10.5 months
Population: Patients achieving a CR (including CMR) or PR (including PMR)
Measure: Median (Full Range); unit: months
Arm/Group | Rituximab, Bendamustine Control | Brentuximab Vedotin Plus Rituximab Plus Bendamustine
Number analyzed (Participants) | 11 | 8
months | 3.7 [0.0 to 10.5] | 4.1 [0.0 to 10.1]

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time randomization to death from any cause
Time Frame: Up to 1.5 years
Population: Intent-to-treat analysis set
Measure: Median (Full Range); unit: months
Arm/Group | Rituximab, Bendamustine Control | Brentuximab Vedotin Plus Rituximab Plus Bendamustine
Number analyzed (Participants) | 12 | 13
months | 14.3 [3.9 to 18] | 6.5 [1.9 to 11.9]

6. Secondary Outcome: Number and Severity of Adverse Events (AEs)
Description: All AEs are included in the summaries, unless treatment-emergent is specified.
Time Frame: Approximately 1 year
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab, Bendamustine Control | Brentuximab Vedotin Plus Rituximab Plus Bendamustine
Number analyzed (Participants) | 12 | 13
Participants
  Treatment-Emergent Adverse Event | 11 | 13
  Treatment-Related Adverse Event | 10 | 13
  Brentuximab Vedotin-Related Adverse Event | 0 | 11
  Rituximab-Related Adverse Event | 6 | 10
  Bendamustine-Related Adverse Event | 10 | 13
  Adverse Event with Outcome of Death | 0 | 1
  Serious Adverse Event | 3 | 8
  Treatment-Related Serious Adverse Event | 3 | 3
  Adverse Event Leading to Dose Delay | 3 | 0
  Adverse Event Leading to Treatment Discontinuation | 1 | 5
  Grade 3-5 Treatment-Emergent Adverse Event | 4 | 11

ADVERSE EVENTS:
Time Frame: 1 year
Description: All AEs (regardless of relationship to study drug) should be recorded from study Day 1 (during and postdose) through the end of the safety reporting period. AE severity is graded using the NCI CTCAE, Version 4.03.
Arm/Group | Rituximab, Bendamustine Control | Brentuximab Vedotin Plus Rituximab Plus Bendamustine
All-Cause Mortality (participants affected / at risk) | 2/12 | 5/13
Serious Adverse Events (participants affected / at risk) | 3/12 | 8/13
Other Adverse Events (participants affected / at risk) | 11/12 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab, Bendamustine Control (N=12) | Brentuximab Vedotin Plus Rituximab Plus Bendamustine (N=13)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Lymphangitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma refractory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (2)
White blood cell count decreased (Investigations) | 0 (0) | 1 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab, Bendamustine Control (N=12) | Brentuximab Vedotin Plus Rituximab Plus Bendamustine (N=13)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 6 (9)
Nausea (Gastrointestinal disorders) | 3 (3) | 5 (7)
Vomiting (Gastrointestinal disorders) | 1 (1) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (6) | 3 (3)
Fatigue (General disorders) | 2 (2) | 3 (6)
Pyrexia (General disorders) | 1 (4) | 4 (5)
Chills (General disorders) | 2 (3) | 0 (0)
Device malfunction (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Performance status decreased (General disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 3 (9) | 1 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 2 (3)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oral fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 2 (6)
Platelet count decreased (Investigations) | 1 (7) | 1 (8)
White blood cell count decreased (Investigations) | 0 (0) | 2 (8)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (2)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (6)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (9)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma refractory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-07-13): https://cdn.clinicaltrials.gov/large-docs/63/NCT02594163/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT02594163/SAP_001.pdf